CLINICAL TRIAL: NCT00958997
Title: Quantitative PET Imaging of Pancreatic Beta-cell Mass in Healthy and Type 1 Diabetic Patients With 18F-FP-DTBZ (AV-133)
Brief Title: Positron Emission Tomography (PET) Imaging of Pancreatic Beta-Cell Mass in Healthy and Type 1 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry); Avid Radiopharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gary Cline, Associate Professor, Yale University
Other Study IDs: Y-003-09
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; islet; pancreas; beta cell mass; PET imaging; FPDTBZ; arginine stimulus test
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — florbenazine F 18; Arginine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 diabetic subjects: Patients with Type 1 diabetes who have a diagnosis of Type 1 diabetes mellitus defined by ADA criteria or judgment of physician
  Interventions: Drug: 18F-FP-DTBZ (18F-AV-133); Biological: Arginine-hydrochloride
- Healthy control subjects: Age-weight-BMI matched to the subjects with type-1 diabetes
  Interventions: Drug: 18F-FP-DTBZ (18F-AV-133); Biological: Arginine-hydrochloride

INTERVENTIONS:
Drug: 18F-FP-DTBZ (18F-AV-133) — The subjects will receive a single IV bolus of approximately 10 mCi 18F-AV-133.(Injection will contain no more than 25 µg of non-radiolabeled 19F-AV-133).
Biological: Arginine-hydrochloride — A bolus injection of 5g of 10% arginine-hydrochloride will be given over a period of 1 minute.

SUMMARY:
Pancreatic Islet beta-cells are responsible for synthesizing and secreting appropriate amounts of insulin to regulate blood glucose levels. One factor in the development of diabetes is the loss of beta-cells. Developing treatments to prevent or restore islet beta-cell mass (BCM) in diabetic patients is hampered by a lack of methods for the non-invasive imaging of these cells. This study is designed to evaluate a radiolabeled compound that binds to the pancreatic islet. The investigators will test the ability of one promising imaging compound, 18F-9-fluoropropyl-(+)-dihydrotetrabenazine (18F-FP-DTBZ), to measure the amount of pancreatic islet beta-cells in patients with long-standing type-1 diabetes and in age-weight-matched healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 1 diabetes may be enrolled if they meet all of the following criteria:

   * Have a diagnosis of Type 1 diabetes mellitus defined by ADA criteria or judgment of physician; diabetes onset younger than age 18, duration >5 years
   * Have fasting C-Peptide ≤ 0.1 ng/ml
   * BMI between 18 and 29 kg/m2
   * Able to tolerate PET and MR imaging
   * No metal implants
   * No claustrophobia
2. Healthy volunteers may be enrolled if they meeting all of the following criteria:

   * Have no history of Type 1 diabetes
   * Fasting blood glucose ≤ 100 mg/dL
   * Negative islet autoantibody testing
   * BMI between 18 and 29 kg/m2
   * Able to tolerate PET and MR imaging
   * No history of previous allergic reactions to drugs
   * No metal implants
   * No claustrophobia

Exclusion Criteria:

* Clinically significant renal dysfunction;
* Clinically significant liver dysfunction as determined by history, physical examination, and standard liver function testing at screening (AST, ALT, Total/Direct Bilirubin, Alkaline Phosphatase);
* Coagulopathy;
* History of allergic reactions to any drug
* Current use of any medications except for insulin for Type 1 diabetes
* Clinically significant cardiovascular disease or clinically significant abnormalities on screening ECG (including but not limited to QTc>450 msec);
* Clinically significant psychiatric disease; Clinically significant pulmonary, renal or hepatic impairment or cancer, have clinically significant infectious disease, including AIDS or HIV infection, or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2; subjects will be asked about this. No testing will be performed.
* Have a history of alcohol or substance abuse or dependence;
* Are women of childbearing potential not refraining from sexual activity or not using adequate contraception. Women must not be pregnant (negative serum β-HCG at the time of screen) or lactating at screening, and must agree to take appropriate steps not to become pregnant during the study and for 30 days following the study.
* Currently receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days.
* Have received a diagnostic or therapeutic radiopharmaceutical within 7 days prior to participation in this study.
* Claustrophobia
* Metal implants (pace-maker, artificial joints, non-removable body piercings)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
PET-determined pancreatic islet beta-cell mass | 150 minutes post-dose of imaging agent

SECONDARY OUTCOMES:
Insulin secretion response following an acute arginine-stimulus test | Six minutes following administration of arginine challange

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Cline, Ph.D., Principal Investigator — Yale University; Yu-Shin Ding, Ph.D., Study Director — Yale University; Kitt F Petersen, M.D., Study Director — Yale University; Richard Carson, Ph.D., Study Director — Yale University
Locations (1):
- Yale University School of Medicine, PET Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Goswami R, Ponde DE, Kung MP, Hou C, Kilbourn MR, Kung HF. Fluoroalkyl derivatives of dihydrotetrabenazine as positron emission tomography imaging agents targeting vesicular monoamine transporters. Nucl Med Biol. 2006 Aug;33(6):685-94. doi: 10.1016/j.nucmedbio.2006.05.006. PMID 16934687
- [Background] Kilbourn MR, Hockley B, Lee L, Hou C, Goswami R, Ponde DE, Kung MP, Kung HF. Pharmacokinetics of [(18)F]fluoroalkyl derivatives of dihydrotetrabenazine in rat and monkey brain. Nucl Med Biol. 2007 Apr;34(3):233-7. doi: 10.1016/j.nucmedbio.2007.01.007. PMID 17383572
- [Background] Kung MP, Hou C, Goswami R, Ponde DE, Kilbourn MR, Kung HF. Characterization of optically resolved 9-fluoropropyl-dihydrotetrabenazine as a potential PET imaging agent targeting vesicular monoamine transporters. Nucl Med Biol. 2007 Apr;34(3):239-46. doi: 10.1016/j.nucmedbio.2006.12.005. PMID 17383573
- [Background] Kung MP, Hou C, Lieberman BP, Oya S, Ponde DE, Blankemeyer E, Skovronsky D, Kilbourn MR, Kung HF. In vivo imaging of beta-cell mass in rats using 18F-FP-(+)-DTBZ: a potential PET ligand for studying diabetes mellitus. J Nucl Med. 2008 Jul;49(7):1171-6. doi: 10.2967/jnumed.108.051680. Epub 2008 Jun 13. PMID 18552132
- [Background] Larsson H, Ahren B. Glucose-dependent arginine stimulation test for characterization of islet function: studies on reproducibility and priming effect of arginine. Diabetologia. 1998 Jul;41(7):772-7. doi: 10.1007/s001250050986. PMID 9686917
- [Background] Rickels MR, Naji A, Teff KL. Acute insulin responses to glucose and arginine as predictors of beta-cell secretory capacity in human islet transplantation. Transplantation. 2007 Nov 27;84(10):1357-60. doi: 10.1097/01.tp.0000287595.16442.a7. PMID 18049122
- [Background] Souza F, Simpson N, Raffo A, Saxena C, Maffei A, Hardy M, Kilbourn M, Goland R, Leibel R, Mann JJ, Van Heertum R, Harris PE. Longitudinal noninvasive PET-based beta cell mass estimates in a spontaneous diabetes rat model. J Clin Invest. 2006 Jun;116(6):1506-13. doi: 10.1172/JCI27645. Epub 2006 May 18. PMID 16710474